CLINICAL TRIAL: NCT05906992
Title: A Double-blind, Randomized, Active-controlled, Parallel Group, Phase 1/3 Study to Compare Efficacy, Pharmacokinetics, Pharmacodynamics and Safety of CT-P53 and Ocrevus in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: A Study to Compare Efficacy, Pharmacokinetics, Pharmacodynamics and Safety of CT-P53 and Ocrevus in Patients With Relapsing-remitting Multiple Sclerosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P53 3.1
Record Dates: First submitted 2023-05-09; First posted 2023-06-18 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- CT-P53 (Experimental): CT-P53(Ocrelizumab)
  Interventions: Biological: CT-P53
- US-Ocrevus (Active Comparator): US-licensed Ocrevus(Ocrelizumab)
  Interventions: Biological: US-Ocrevus
- EU-Ocrevus (Active Comparator): EU-approved Ocrevus(Ocrelizumab)
  Interventions: Biological: EU-Ocrevus

INTERVENTIONS:
Biological: CT-P53 — Intravenous(IV) infusion
  Other Names: Ocrelizumab
  Arms: CT-P53
Biological: US-Ocrevus — Intravenous(IV) infusion
  Other Names: Ocrelizumab
  Arms: US-Ocrevus
Biological: EU-Ocrevus — Intravenous(IV) infusion
  Other Names: Ocrelizumab
  Arms: EU-Ocrevus

SUMMARY:
This is a double-blind, randomized, active-controlled, parallel group, Phase 1/3 study to compare efficacy, PK, PD and overall safety of CT-P53 with Ocrevus in patients with Relapsing-remitting Multiple Sclerosis.

DETAILED DESCRIPTION:
CT-P53, containing the active ingredient ocrelizumab, is a humanized monoclonal antibody that is being developed as a proposed biosimilar medicinal product to Ocrevus. The purpose of this study is to demonstrate similar efficacy, PK, PD and safety of CT-P53 and Ocrevus in patients with Relpasing-remitting Multiple Screlosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed as multiple sclerosis (MS) in accordance with the revised McDonald criteria.
* Patient has evidence of recent MS activity as defined in the study protocol
* Patient has neurological stability for ≥30 days.
* Patient with 0 to 6.0 (both inclusive) on the EDSS score.

Exclusion Criteria:

* Patient diagnosed with primary or secondary progressive MS.
* Patient diagnosed with MS for more than 15 years duration with an EDSS score ≤2.0 at Screening.
* Patient unable to complete or has a contraindication to an MRI
* Patient with contraindications and/or severe hypersensitivity to corticosteroids including methylprednisolone or any of the excipients of study drug or etcs defined in the study protocol.
* Patient who has currently or history of any of medical conditions described in the study protocol.
* Patients who have received or going to receive any of prohibited medications or treatments defined in the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 512 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve in PK group | Up to Week 24
  To demonstrate PK comparability in terms of the area under the concentration time curve in patients with RRMS as follows:
  * Area under the concentration-time curve from time zero to Week 2 (AUC0-wk2)
  * Area under the concentration-time curve from Week 2 to Week 24 (AUCwk2-wk24)
Total number of new GdE lesions on T1-weighted brain MRI in Main study group | Up to Week 24
  To demonstrate the equivalence of CT-P53 to reference drug (EU-Ocrevus and US-Ocrevus) in terms of efficacy in patients with RRMS as determined by the total number of new gadolinium-enhancing (GdE) lesions on T1-weighted brain magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Absoulte CD19+ B-cell counts for PD assessments | Up to Week 96
  To assess PD of CT-P53 and reference drug (EU-Ocrevus and US-Ocrevus) as follows:
  • Absolute CD19+ B-cell counts
Area under the concentration-time curve in PK group | Up to Week 16
  Area under the concentration-time curve from time zero to Week 16
Total body clearance in PK group | Up to Week 2
  Total body clearance covering both administrations at Weeks 0 and 2 (CL)
Volume of distribution at steady state in PK group | Up to Week 2
  Volume of distribution at steady state covering both administrations at Week 0 and 2 (Vss)
Safety: Immunogenecity | Up to Week 96
  Number and percentage of patients with positive antidrug-antibody and neutralizing antibody results
Annualized Relapse Rate (ARR) | Up to Week 96
  The total number of protocol-defined MS relapses for each patient will be counted and listed. Annualized relapse rate (ARR) will be calculated by the total number of protocol-defined relapses for all patients divided by time-in-study by patient.
Change in Expanded Disability Status Score (EDSS) | Up to Week 96
  The EDSS score will be listed and descriptive statistics for actual value and change in EDSS score from baseline to Weeks 24, 48 and 96 will be summarized by treatment group and visit.
  An increase ≥1.5 point from baseline EDSS score is defined as disability progression.
  A reduction ≥1.0 point from baseline EDSS score is defined as disability improvement.
Change in Multiple Sclerosis Functional Composite Score (MSFCS) | Up to Week 96
  There are three components to the MSFCS; (1) the average scores of two trials of T25-FW (2) the average scores on the 9-HPT (the two trials for each hand are averaged, converted to the reciprocals of the mean times for each hand and then the two reciprocals are averaged) (3) the number of correct answers from the PASAT-3. Multiple Sclerosis Functional Composite Score (MSFCS) is based on the concept that scores for these three dimensions (arm, leg, and cognitive functions) are combined to create a single score (the MSFCS) that can be used to detect change over time in MS patients
Total Number of Lesions on Brain Magnetic Resonance Imaging | Up to Week 96
  The total number of lesions on brain MRI will be calculated as the cumulative sum of the individual number of the lesions at each scheduled visit
Volume of Hypointense Lesions on T1-weighted Brain Magnetic Resonance Imaging | Up to Week 96
  Actual value of volume of hypointense lesions on T1-weighted brain MRI will be listed by treatment group and visit. Descriptive statistics for actual value and change in volume of hypointense lesions on T1-weighted brain MRI from baseline to Weeks 24, 48 and 96 will be summarized by treatment group
Brain Volume on Brain Magnetic Resonance Imaging | Up to Week 96
  Change in brain volume is defined as the brain volume at pre-specified time point minus brain volume at baseline. Actual value of brain volume on brain MRI will be listed by treatment group. Descriptive statistics for actual value and percentage change in brain volume on brain MRI from baseline to Weeks 24, 48 and 96 will be summarized by treatment group.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to Week 96
  All reported terms of AEs will be coded to system organ class (SOC) and preferred term (PT) according to the Medical Dictionary for Regulatory Activities (MedDRA) and severity grading of AEs will be recorded according to the CTCAE Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Minji Ma, Study Chair — Celltrion, Inc.
Locations (1):
- CT-P53 3.1 investigational site, Poznan, Poland